CLINICAL TRIAL: NCT05701800
Title: A Phase 1/2, Randomized, Observer-Blind, Active-Controlled, Dose-Ranging Study to Evaluate the Safety, Reactogenicity and Immunogenicity of mRNA-1468, a Candidate Vaccine to Prevent Herpes Zoster (HZ) in Healthy Adults ≥50 Years of Age
Brief Title: A Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1468 in Healthy Adults ≥50 Years of Age
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: mRNA-1468-P101
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Herpes Zoster
Keywords: mRNA-1468; Herpes Zoster vaccine; Moderna
MeSH Terms: conditions — Herpes Zoster | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1: mRNA-1468: Dose 1 (Experimental): Participants will receive placebo by intramuscular (IM) injection on Day 1 followed with mRNA-1468 by IM injection on Day 57 in Part 1.
  Interventions: Biological: mRNA-1468; Biological: Placebo
- Part 1: mRNA-1468: Dose 2 (Experimental): Participants will receive mRNA-1468 by IM injection on Day 1 and Day 57 in Part 1.
  Interventions: Biological: mRNA-1468
- Part 1: mRNA-1468: Dose 3 (Experimental): Participants will receive mRNA-1468 by IM injection on Day 1 and Day 57 in Part 1.
  Interventions: Biological: mRNA-1468
- Part 1: mRNA-1468: Dose 4 (Experimental): Participants will receive mRNA-1468 by IM injection on Day 1 and Day 57 in Part 1.
  Interventions: Biological: mRNA-1468
- Part 1: Shingrix (Active Comparator): Participants will receive Shingrix by IM injection on Day 1 and Day 57 in Part 1.
  Interventions: Biological: Shingrix
- Part 2: mRNA-1468: Dose 5 (Experimental): Participants will receive mRNA-1468 by IM injection on Day 1 and Day 57 in Part 2.
  Interventions: Biological: mRNA-1468
- Part 2: mRNA-1468: Dose 6 (Experimental): Participants will receive mRNA-1468 by IM injection on Day 1 and Day 57 in Part 2.
  Interventions: Biological: mRNA-1468
- Part 2: Shingrix (Active Comparator): Participants will receive Shingrix by IM injection on Day 1 and Day 57 in Part 2.
  Interventions: Biological: Shingrix

INTERVENTIONS:
Biological: mRNA-1468 — Sterile liquid dispersion for injection
  Arms: Part 1: mRNA-1468: Dose 1; Part 1: mRNA-1468: Dose 2; Part 1: mRNA-1468: Dose 3; Part 1: mRNA-1468: Dose 4; Part 2: mRNA-1468: Dose 5; Part 2: mRNA-1468: Dose 6
Biological: Placebo — Sterile liquid for injection
  Other Names: Saline
  Arms: Part 1: mRNA-1468: Dose 1
Biological: Shingrix — Sterile suspension for injection
  Arms: Part 1: Shingrix; Part 2: Shingrix

SUMMARY:
The purpose of this first-in-human study is to evaluate the safety and immunogenicity of mRNA-1468.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Is an adult 50 years of age or older at the time of consent. Part 2: Is an adult 50-69 years of age at the time of consent.
* Has a body mass index of 18 to <40 kilograms/meter squared at the Screening Visit.
* Females of childbearing potential: have a negative pregnancy test at the Screening Visit and on the day of the first vaccination (Day 1); have practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1; have agreed to continue adequate contraception through 3 months following vaccine administration; are not currently breastfeeding.

Exclusion Criteria:

* Has a history of HZ within the past 10 years.
* Has been previously vaccinated against varicella or HZ.
* Is acutely ill or febrile
* Body temperature ≥38.0°Celsius/100.4°Fahrenheit 72 hours prior to or at the Screening Visit or on Day 1. Participants meeting this criterion may be rescheduled within the allowed window.
* Has a current or previous diagnosis of congenital or acquired immunodeficiency, immunocompromizing/immunosuppressive condition, asplenia, or recurrent severe infections. Certain immune-mediated conditions that are well controlled and stable (for example, Hashimoto thyroiditis) as well as those that do not require systemic immunosuppressive therapy (for example, asthma, psoriasis, or vitiligo) may be permitted at the discretion of the Investigator.
* Has a dermatologic condition that could affect local solicited adverse reaction assessments (for example, tattoos, psoriasis patches affecting skin over the deltoid areas).
* Has any medical, psychiatric, or occupational condition, including reported history of substance abuse, that, in the opinion of the Investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.
* Has a history of myocarditis, pericarditis, or myopericarditis.
* Has a reported history of anaphylaxis or severe hypersensitivity reaction after receipt of any mRNA vaccine(s) or any components of the mRNA vaccines.
* Has received systemic immunosuppressants for >14 days in total within 180 days prior to Screening Visit (for corticosteroids ≥10 milligrams/day of prednisone or equivalent) or is anticipating the need for systemic immunosuppressive treatment at any time during participation in the study. Inhaled, nasal, intra-articular and topical steroids are allowed.
* Has received systemic immunoglobulins, long-acting biological therapies that affect immune responses (for example, Infliximab) or blood products within 90 days prior to the Screening Visit or plans to receive them during the study.

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 659 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number Participants with Solicited Local and Systemic Reactogenicity Adverse Reactions | Up to Day 64 (7 days after each injection)
Number of Participants with Unsolicited Adverse Events (AEs) | Up to Day 85 (28 days after each injection)
Number of Participants with Serious AEs, AEs Leading to Discontinuation of Study Vaccine or Withdrawal From the Study, and AEs of Special Interest | Day 1 to End of Study (up to a maximum of Day 1113)
Number of Participants with Medically Attended AEs | Day 1 to Day 393 (12 months after last study injection)

SECONDARY OUTCOMES:
Vaccine Seroresponse Rate of Participants | Day 85 and Day 225 (1 and 6 months after the last injection)
  Vaccine seroresponse will be defined as an anti-glycoprotein E (gE)-specific binding antibody (bAb) concentration ≥4-fold if baseline bAb concentration is above the lower limit of quantification (LLOQ) or ≥4 * LLOQ if baseline bAb concentration is <LLOQ prior to vaccination.
Geometric Mean Concentration of Anti-gE-specific bAb as Measured by Enzyme-linked Immunosorbent Assay | Day 85 and Day 225 (1 and 6 months after the last injection)
Change from Baseline in Geometric Mean Fold Rise of Anti-gE-specific bAb Concentration | Baseline, Day 85 and Day 225 (1 and 6 months after the last injection)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (19):
  - Velocity Clinical Research - Westlake, Los Angeles, California
  - Tekton Research, Inc - Longmont Center, Longmont, Colorado
  - Meridien Research, Lakeland, Florida
  - Clinical Trials of Florida, LLC, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Florida Pulmonary Research Institute, LLC, Winter Park, Florida
  - Centricity Research, Columbus, Georgia
  - Great Lakes, Chicago, Illinois
  - DM Clinical Research- River Forest, River Forest, Illinois
  - Meridian Clinical Research - Dakota Dunes, Sioux City, Iowa
  - Johnson County Clin-Trials (JCCT), Lenexa, Kansas
  - NOLA Research Works, New Orleans, Louisiana
  - Velocity Clinical Research - Medford, Medford, Oregon
  - DM Clinical Research - Philadelphia, Philadelphia, Pennsylvania
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Tekton Research, Austin, Texas
  - Gadolin Research, Beaumont, Texas
  - LinQ Research, LLC, Houston, Texas
  - DM Clinical Research, Tomball, Texas
- Research Works San Juan, San Juan, Puerto Rico